CLINICAL TRIAL: NCT03264378
Title: Partnership in Implementation Science for Geriatric Mental Health (PRISM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Society and Health Institute (Thailand) (Unknown); Shanghai Mental Health Center (China) (Unknown); University of South Carolina (Other); University of California, Davis (Other)
Responsible Party: Principal Investigator, Hongtu Chen, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2017P000186/PHS
Record Dates: First submitted 2017-08-24; First posted 2017-08-29 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Behavioral and Psychological Symptoms of Dementia (BPSD)
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: The experimental group will receive physical exercise intervention (PEI) that is supported by standardized administrative procedures plus the GTO-ThAI implementation support system designed to improve the quality of implementation of the PEI program. The active comparator group will receive PEI that is supported only by standardized administrative procedures that the Thai government typically uses to promote policy-driven initiatives.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: None of participants, care providers, or outcome assessor knows whether which participants have been assigned to intervention or control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEI-GTO-ThAI (Experimental): Physical exercise intervention (PEI) supported by the GTO-ThAI Implementation Model
  Interventions: Behavioral: Physical Exercise Intervention
- PEI-Standard (Active Comparator): Physical exercise intervention (PEI) supported by the standard governmental administrative procedures
  Interventions: Behavioral: Physical Exercise Intervention

INTERVENTIONS:
Behavioral: Physical Exercise Intervention — The 12-week physical exercise intervention will be delivered by trained community health workers (CHW) who are supervised by nurses. The CHW will visit the patient's home-3 sessions per week for the first 2 weeks, followed by weekly visits for 6 weeks, and then weekly telephone support for 4 weeks-to instruct the family caregiver and the patient in the exercise routine. Each session includes physical activities designed to promote gentle stretching, strength, balance, flexibility, and endurance, with a progressive schedule (i.e., the total length of time increases from 10 minutes up to 30 minutes maximum) and its intensity adjusted based on the participant's level of fitness.

SUMMARY:
The Partnership in Implementation Science for Geriatric Mental Health (PRISM) project proposes an evidence-based physical exercise intervention for older adults who exhibit behavioral and psychological symptoms of dementia (BPSD). The proposed evaluation study will conduct a randomized controlled trial with a Hybrid Type 3 design to compare the intervention arm that implements the culturally-adapted GTO model (GTO-ThAI) to deliver implementation support, with a control arm, which receives usual top-down administrative instruction for implementing a policy initiative.

DETAILED DESCRIPTION:
The overall goal of this project is to establish a hub to integrate implementation research for scaling up sustainable, evidence-based mental health interventions with research capacity-building activities for East Asia. Specific scale-up study aims include: Aim 1: Assessing readiness for implementing the evidence-based physical exercise intervention for improving mental health of older adults in participating provinces of Thailand; Aim 2: Developing the GTO-ThAI implementation support model through a pre-implementation case study and formative evaluation; and Aim 3: Evaluation of implementation strategies and clinical outcomes through a hybrid Type 3 randomized trial to test an evidence-based implementation support strategy (i.e., the GTO-ThAI model) that emphasizes a systematic process to address implementation barriers to the delivery of the evidence-based physical exercise intervention (PEI), compared with the existing standard administrative procedures for delivering the same PEI.

ELIGIBILITY:
Inclusion Criteria:

* (a) adults who are aged 55 and older,
* (b) screen positive for dementia,
* (c) screen positive for BPSD, and
* (d) having a caregiver who is willing to participate in the study.

Exclusion Criteria:

* (a) caregivers who are cognitively not intact, and/or
* (b) not willing to participate in the intervention.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Implementation outcome score | Up to 12 months
  Adapted from the Quality Implementation Tool (Meyer et al., 2012), using a total score based on average of ratings, by site implementation team leaders, on a 7-point Likert scale over 48 items across eight dimensions of implementation (e.g. adoption, fidelity, dosage, program reach, differentiation, quality of implementation, implementation cost, sustainability).

SECONDARY OUTCOMES:
Behavioral and psychological symptoms of dementia (BPSD) | Up to 12 months
  BPSD will be assessed by the Neuropsychiatric Inventory (NPI), using the total score obtained by summing all the individual domain total scores; each domain score is the product of the frequency score multiplied by the severity score for that behavioral domain.

CONTACTS AND LOCATIONS:
Overall Officials: Hongtu Chen, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Ministry of Public Health, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
We don't have a plan to share individual participant data.

REFERENCES:
- [Derived] Chen H, Levkoff S, Chuengsatiansup K, Sihapark S, Hinton L, Gallagher-Thompson D, Tongsiri S, Wisetpholchai B, Fritz S, Lamont A, Domlyn A, Wandersman A, Marques AH. Implementation Science in Thailand: Design and Methods of a Geriatric Mental Health Cluster-Randomized Trial. Psychiatr Serv. 2022 Jan 1;73(1):83-91. doi: 10.1176/appi.ps.202000028. Epub 2021 Jun 15. PMID 34126778